CLINICAL TRIAL: NCT05761132
Title: Neo-adjuvant Pembrolizumab in Vulvar Squamous Cell Carcinoma: a Clinical Proof-of-concept Study
Acronym: Apollo
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: University Medical Center Groningen (Other); Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Mariette I. E. van Poelgeest, Principle Investigator, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Apollo
Record Dates: First submitted 2022-08-11; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Vulva Cancer; Vulva Neoplasm; Squamous Cell Cancer
Keywords: pembrolizumab; immunotherapy; neoadjuvant
MeSH Terms: conditions — Vulvar Neoplasms; Neoplasms, Squamous Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Neoadjuvant pembrolizumab (Experimental): Patients receive pembrolizumab, 200 mg IV Q3W for a total of 2 administrations per patient over a period of 6 weeks prior to surgery.
  Responders have the option to fall into an extension cohort and, after consultation with the multidisciplinary team, will be treated with adjuvant pembrolizumab from week 16 until week 58 (400 mg IV, Q6W, 7 times).
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — neoadjuvant immunotherapy
  Other Names: checkpoint inhibitor

SUMMARY:
Rationale:

Vulvar squamous cell carcinoma (VSCC) is a rare cancer with a rising incidence. Standard treatment comprises wide local excision of the primary tumour and inguinal lymph nodes and sometimes (chemo) radiotherapy. Treatment is associated with impressive and long-lasting morbidity, sexual and psychological dysfunction and wound healing disorders. Recurrent disease develops in up to 40% of all treated patients. The unmet need, therefore, is a less radical and more effective treatment for VSCC.

Hypothesis:

Based on the local immune profile in a large fraction of patients with primary VSCC the investigators hypothesize that neoadjuvant PD-1 checkpoint inhibition may reinvigorate tumor-specific T cells resulting in a reduced tumor load, potentially leading to less radical surgery and reduces the recurrence rate.

The primary objectives of this trial are to study clinical efficacy and immune activation of neoadjuvant PD-1 blockade in VSCC.

Study design: This is a prospective, multicenter phase II non-controlled clinical trial in 40 VSCC patients.

Study population: Clinically diagnosed FIGO I-III primary VSCC patients to be treated with surgery with curative intent.

Intervention (if applicable):

Anti-PD1 antibody pembrolizumab, 200 mg IV Q3W for a total of 2 administrations per patient over a period of 6 weeks prior to surgery.

Main study parameters/endpoints:

The primary endpoints are:

* Clinical efficacy of neoadjuvant PD-1 blockade in VSCC, measured by objective change in tumour size (according to RECIST1.1)
* The activation, proliferation and migration of the CD4+CD39+PD-1+ intratumoral T-cell population.

DETAILED DESCRIPTION:
Rationale:

Vulvar squamous cell carcinoma (VSCC) is a rare cancer with a rising incidence. Standard treatment comprises wide local excision of the primary tumour and inguinal lymph nodes and sometimes (chemo) radiotherapy. Treatment is associated with impressive and long-lasting morbidity, sexual and psychological dysfunction and wound healing disorders. Recurrent disease develops in up to 40% of all treated patients. The unmet need, therefore, is a less radical and more effective treatment for VSCC.

Hypothesis:

Based on the local immune profile in a large fraction of patients with primary VSCC the investigators hypothesize that neoadjuvant programmed cell death protein 1 (PD-1) checkpoint inhibition may reinvigorate tumor-specific T cells resulting in a reduced tumor load, potentially leading to less radical surgery and reduces the recurrence rate.

The primary objectives of this trial are to study clinical efficacy and immune activation of neoadjuvant PD-1 blockade in VSCC.

Study design: This is a prospective, multicenter phase II non-controlled clinical trial in 40 VSCC patients.

Study population: Clinically diagnosed FIGO I-III primary VSCC patients to be treated with surgery with curative intent.

Intervention (if applicable):

Anti-PD1 antibody pembrolizumab, 200 mg IV Q3W for a total of 2 administrations per patient over a period of 6 weeks prior to surgery.

Main study parameters/endpoints:

The primary endpoints are:

* Clinical efficacy of neoadjuvant PD-1 blockade in VSCC, measured by objective change in tumour size (according to RECIST1.1)
* The activation, proliferation and migration of the CD4+CD39+PD-1+ intratumoral T-cell population.

The secondary endpoints are:

* Pathological complete responses (pCR) at time of surgery
* Feasibility (defined as delay in planned surgery and surgical outcomes), safety according to NCI-CTC version 5.0,
* The activation, proliferation and migration of the CD8+CD103+CD39+PD-1+ intratumoral T-cell population upon PD-1 blockade.

Exploratory endpoints:

* To study the on-treatment effect of neoadjuvant PD-1 blockade on a) Local RNA-based immune signalling; b) The activation, proliferation and migration of CD39-negative T cells; c)The type 1 cytokine polarization of T cells as indicated by the percentage of Tbet+ T cells; d) The myeloid cell component, as determined by multiplex staining for CD68, CD14, CD11c, CD33, HLA-DR and CD163, present in VSCC tumors.
* To study the relation between the T-cell inflamed gene expression profile (GEP) score and PD-1 blockade driven immunological changes in the tumor microenvironment (TME).
* To study the relation between the T-cell infiltration pattern and PD-1 blockade driven immunological changes in TME.
* To study the relation between immune cell changes in the TME and corresponding immune cells in the blood.
* To study immune cell composition in TME post neoadjuvant checkpoint blockade by AURORA flow cytometry on fresh resection material.
* To study PD-L1 expression and molecular subtype (HPV+, p53mut, other) in tumor material.
* To assess quality of life (EORTC QLQ C-30 and QLQ-VU34).
* To study the utility of plasma-derived circulating tumor DNA (ctDNA) as a potential future predictor for minimal residual disease and/or relapse.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow-up assessments.
2. Age ≥ 18 years old at the day of signing informed consent
3. Histologically confirmed primary vulvar squamous cell carcinoma, with all of the following characteristics:

   * At least 1 lesion that can be measured in at least 1 dimension with ≥ 10 mm in largest diameter.
   * Clinically stage FIGO I-III.
   * Documentation confirming the absence of distant metastasis (M0) as determined by institutional practice. Routine exams to discard metastases will be performed according to Investigator judgement but are mandatory in case of suspicion of metastatic disease.
   * Vulvar cancer eligible for primary surgery
   * In the case of a multifocal tumor (defined as the presence of two or more foci of cancer on the vulva), the largest lesion must be ≥ 10 mm and all lesions ≥ 10 mm are designated as "target" lesion(s) for all subsequent tumor evaluations and biopsies.
4. ECOG performance 0-1
5. Have adequate organ function as measured within 28 days prior to administration of study treatment.
6. A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

   * Is not a woman of childbearing potential, or
   * Is a woman of childbearing potential and using a contraceptive method that is highly effective (with a failure rate of <1% per year), with low user dependency, or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis), as described in Appendix 11 during the intervention period and for at least the time needed to eliminate each study intervention after the last dose of study intervention and agrees not to donate eggs (ova, oocytes) to others or freeze/store for her own use for the purpose of reproduction during this period. The length of time required to continue contraception for each study intervention is 120 days for pembrolizumab.

Exclusion Criteria:

1. Locally advanced tumor not amenable to surgical therapy.
2. A woman of child bearing potential who has a positive urine pregnancy test within 72 hours prior to allocation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
3. Prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD37)
4. Prior systemic anti-cancer therapy including investigational agents within 4 weeks [prior to allocation.

   Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible.

   Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
5. Prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
6. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
7. A live vaccine within 30 days before the first dose of study intervention. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette- Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed. Please refer to section 5.4 for information on COVID-19 vaccines.
8. Currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment. Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
9. Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
10. A known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin on a location other than the vulva, or carcinoma in situ (e.g. of the breast , cervix or bladder) that have undergone potentially curative therapy are not excluded.
11. Severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
12. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    * Patients with vitiligo or alopecia
    * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    * Any chronic skin condition that does not require systemic therapy
    * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
    * Patients with celiac disease controlled by diet alone
13. History of (non-infectious) pneumonitis that required steroids or has current pneumonitis
14. An active infection requiring systemic therapy.
15. Known history of Human Immunodeficiency Virus (HIV). Note: No HIV testing is required unless mandated by local health authority.
16. Known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
17. A history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the subject's participation for the full duration of the study in such it is not in the best interest of the subject to participate, in the opinion of the treating investigator.
18. Is pregnant or breastfeeding or expecting to conceive within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
19. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
20. Has had an allogenic tissue/solid organ transplant.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
objective response rate (according to RECIST1.1) | 6 weeks
  reponse rate
The numbers of CD4+CD39+ T cells expressing PD-1+ and/or HLA-DR+ with or without co-expression of ki67 (per m2 stroma and tumor) | 6 months
  activation, proliferation and migration of the CD4+CD39+PD-1+ intratumoral T-cell population; PD

SECONDARY OUTCOMES:
Pathological complete responses | 8 weeks
  pCR
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 3 months
  Toxicity (according to NCI-CTC v5)
The number of intratumoral CD8+CD103+CD39+PD-1+ T-cell population upon PD-1 blockade | 6 months
  PD

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Poelgeest MIE, Kortekaas KE, van Doorn HC, Oonk M, Nijman HW, Boere I, Eerkens AL, Reyners AKL, Ewing-Graham PC, Bart J, Bosse T, Welters MJP, Kroep JR, van der Burg SH. APOLLO: neo-adjuvant pembrolizumab for primary vulvar squamous cell carcinoma-a multicenter, single-arm, phase II, clinical proof-of-concept study. Int J Gynecol Cancer. 2025 Oct;35(10):101831. doi: 10.1136/ijgc-2024-005523. Epub 2025 Apr 17. PMID 38909994